CLINICAL TRIAL: NCT01698788
Title: Role of Intraoperative Dexamethasone Implant in Improving Outcome of Taut Posterior Hyaloid Removal in Diabetic Macular Edema
Brief Title: Effect of Intraoperative Dexamethasone Implant in Taut Posterior Hyaloid Removal in Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Pooja Bansal,MD, MD, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: dr.poojabansal
Record Dates: First submitted 2012-03-22; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Diabetic Macular Edema; Vision Disorders
Keywords: diabetic macular edema; taut posterior hyaloid membrane; ozurdex
MeSH Terms: conditions — Vision Disorders | interventions — Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TPHM removal without ozurdex (Experimental): Comparison of taut posterior hyaloid removal with (Group B)and without intraoperative ozurdex(Group A)
  Interventions: Drug: Dexamethasone Drug delivery system (Ozurdex)
- TPHM removal with ozurdex (Experimental): Comparison of TPHM removal with (Group B) and without (Group A)Ozurdex
  Interventions: Drug: Dexamethasone Drug delivery system (Ozurdex)

INTERVENTIONS:
Drug: Dexamethasone Drug delivery system (Ozurdex) — It is a sustained release intravitreal implant containing 700µg dexamethasone
  Other Names: OZURDEX

SUMMARY:
This study is undertaken to determine effect of sustained release dexamethasone implant,Ozurdex in improving outcome of taut posterior hyaloid removal in patients with diabetic macular edema

Diabetic macular edema constitute important cause of visual impairment in patients with diabetes.Focal/ grid laser photocoagulation is the standard of care in the management . Several adjuncts including intravitreal corticosteroids, Pegaptanib Sodium , Ranibizumab , Bevacizumab are also been tried.In some patients inspite of multiple lasers or injections macular edema persists as a consequence overlying taut posterior hyaloid membrane which needs to be removed by vitrectomy. Visual improvement after vitrectomy is related to the duration of edema, as well as the extent of intraretinal lipid and vascular nonperfusion.Even after surgery some patients might need repeat intravitreal bevacizumab or triamcinolone injections to take care of residual macular edema.Intravitreal Triamcinolone Acetonide (TA), a water insoluble steroid, has been shown to reduce the retinal thickness and improve the visual acuity. However, recurrence of macular edema in patients who receive intravitreal TA is a major concern because of its short half life . In search for the ideal corticosteroid preparation, a Dexamethasone Posterior Segment Drug Delivery System (Dexamethasone DDS - Ozurdex®, Allergan Inc, Irvine, California) was recently developed which has generated new interest in this molecule. It is a sustained release intravitreal implant containing 700µg dexamethasone has been approved by the US-FDA (Food and Drug Administration) for treatment of macular edema in retinal vein occlusions. The present study introduces a novel concept of using intraoperative Ozurdex ® implant during taut posterior hyaloid removal and its effect in improving the surgical outcome

DETAILED DESCRIPTION:
This study is undertaken to determine effect of sustained release dexamethasone implant,Ozurdex in improving outcome of taut posterior hyaloid removal in patients with diabetic macular edema

Diabetic macular edema constitute important cause of visual impairment in patients with diabetes.Focal/ grid laser photocoagulation is the standard of care in the management .Several adjuncts including intravitreal corticosteroids, Pegaptanib Sodium , Ranibizumab , Bevacizumab are also been tried.In some patients inspite of multiple lasers or injections macular edema persists as a consequence overlying taut posterior hyaloid membrane which needs to be removed by vitrectomy. The exact role of vitreous in the pathogenesis of diabetic maculopathy remains unclear although it has been implicated as a cause of macular edema via several mechanical and physiologic mechanisms, which include the following (1) destabilization of the vitreous by abnormal glycation and crosslinking of vitreal collagen, leading to traction on the macula, (2) accumulation and concentration of factors causing vasopermeability in the premacular vitreous gel and (3) accumulation of chemoattractant factors in the vitreous, leading to cellular migration to the posterior hyaloid, contraction and macular traction. The observation that release of mechanical traction on the macula with subsequent reduction in DME, either by spontaneous posterior vitreous detachment or with vitrectomy, lends support to this line of reasoning. Furthermore, the evidence that vitrectomy produces improved retinal oxygenation taken together with the evidence that increased oxygenation can reduce DME, suggests an additional physiologic advantage but determination of which eyes might benefit from vitrectomy is the most challenging aspect in the treatment of this condition. Fluorescein angiography, B-scan ultrasonography, and optical coherence tomography may be helpful in this regard. Most often, vitreous surgery is performed when diabetic macular edema persists despite multiple laser treatments. All reports published to date regarding vitrectomy for diabetic macular edema are uncontrolled and nonrandomized patient series. Visual improvement after vitrectomy is related to the duration of edema, as well as the extent of intraretinal lipid and vascular nonperfusion.Even after surgery some patients might need repeat intravitreal bevacizumab or triamcinolone injections to take care of residual macular edema.Intravitreal Triamcinolone Acetonide (TA), a water insoluble steroid, has been shown to reduce the retinal thickness and improve the visual acuity. However, recurrence of macular edema in patients who receive intravitreal TA is a major concern because of its short half life . In search for the ideal corticosteroid preparation, a Dexamethasone Posterior Segment Drug Delivery System (Dexamethasone DDS - Ozurdex®, Allergan Inc, Irvine, California) was recently developed which has generated new interest in this molecule. It is a sustained release intravitreal implant containing 700µg dexamethasone has been approved by the US-FDA (Food and Drug Administration) for treatment of macular edema in retinal vein occlusions. The present study introduces a novel concept of using intraoperative Ozurdex ® implant during taut posterior hyaloid removal and its effect in improving the surgical outcome

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or 2 Diabetes mellitus
2. TPHM causing cystoid macular edema with or without subfoveal serous RD on OCT

Exclusion Criteria:

1. Known case of ocular hypertension or glaucoma
2. Macular ischemia on FFA

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
change in central macular thickness | Baseline to 3 months
  The primary outcome measure is the change in the central macular thickness, either an increase or decrease, as measured by optical coherence tomography as compared to the preoperative thickness

SECONDARY OUTCOMES:
change in visual acuity | Baseline to 3 months
  Change in the visual acuity as measured by the logMAR visual acuity chart

CONTACTS AND LOCATIONS:
Overall Officials: POOJA BANSAL, MBBS,MS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; VISHALI R GUPTA, MBBS,MS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; AMOD GUPTA, MBBS,MS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Pooja Bansal, Chandigarh, Chandigarh, India